CLINICAL TRIAL: NCT01753960
Title: Noninvasive and Continuous Hemoglobin Monitoring for Surgical Blood Management (NACHO) - Matched-pair Cluster-randomized Controlled Trial
Brief Title: Surgical Blood Management Using Noninvasive and Continuous Hemoglobin Monitoring(NACHO)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-12-IM-0561-12-CTIL
Record Dates: First submitted 2012-11-05; First posted 2012-12-20 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2013-01

CONDITIONS: Hemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group: Anesthesiologists without access to data from a continuous noninvasive hemoglobin monitoring device during surgery.
- SpHb group: Anesthesiologists with access to data from a continuous noninvasive hemoglobin monitoring device during surgery.

SUMMARY:
The purpose of this study is to determine whether Noninvasive and Continuous Hemoglobin Monitoring (NACHO) for Surgical Blood Management affects transfusion decision making algorithm in the operating room.

DETAILED DESCRIPTION:
Blood transfusions are associated with various risks including viral infections, delayed wound healing, transfusion related acute lung injury and cardiovascular complications. Despite limitations, and ongoing efforts to identify and validate other more-physiologically-relevant "triggers" for blood transfusions, hemoglobin-based transfusion triggers are still commonly used in practice, as well as in all currently available transfusion guidelines, alone, or in combination with other parameters. In the operating room the anesthesiologist has to withdraw blood from the patient and send it to the lab or the blood gas machine to achieve hemoglobin levels. It may be suggested that the ability to continuously monitor hemoglobin levels may help physicians to take more appropriate transfusion decisions; i.e, the physicians will either identify critical decreases in hemoglobin levels earlier and respond appropriately or avoid over-transfusing when hemoglobin levels have not decreased yet. Accordingly, monitors of hemoglobin levels are used in the operating theatre in many centers, although their blood-conserving effect has not been proven yet.

We believe that the transfusion decision making algorithm in the operating room relies less heavily on "on spot" measures of hemoglobin levels but rather on patient's comorbidities, expected additional bleeding according to the surgery and the surgeon, the course of the operation (the operating field is "open" and thus surgeons can tell if it is oozing or frank bleeding, if they can control bleeding promptly or not etc..), hemodynamic data available from the different invasive and non-invasive monitors, pressure from the surgeon, etc. It is therefore suggested that continuous monitoring of hemoglobin levels may be less relevant in this environment.

Specific Aims/Hypothesis:

1. The primary hypothesis is that continuous noninvasive hemoglobin monitoring will not reduce the number of blood transfusions in patients undergoing surgeries associated with a significant risk of bleeding.
2. The secondary hypothesis is that in patients monitored with continuous noninvasive hemoglobin, there will not be earlier warning of critical drops in hemoglobin, resulting in less frequent complications compared with patients who are not being monitored with continuous noninvasive hemoglobin.

ELIGIBILITY:
1. Anesthesiologists Eligibility Criteria

   Inclusion Criteria:
   * Consenting anesthesiologist
   * Anticipate to manage at least 10 cases per month
   * At least 3-year post-graduate clinical experience as an anesthesiologist responsible for making transfusion decisions for individual patients

   Exclusion Criteria:
   * Not meeting the appropriate licensing requirements
   * No being board-certified in Anesthesiology
   * Inability or unwillingness to complete study-related procedures, including undergoing training with regards to using and interpreting the monitor data in the operating room
2. Eligible patients under the case of the consenting eligible Anesthesiologist.

Inclusion criteria:

150 Adult patients undergoing major surgeries associated with possibility of significant blood loss (e.g. such that blood is cross-matched and available before the start of the case as per hospital routine practice).

* Consenting patients who are primarily managed by the consenting anesthesiologists participating in the study
* At least one finger available and accessible for performing non-invasive hemoglobin monitoring.

Exclusion criteria:

* Any patients who do not fit the criteria for use of sensor, specifically, any patient with nail polish and/or a nail deformity, or obstructed physical access (e.g. due to bandage) to all fingers that would be used for sensor placement, in a manner that interferes with satisfactory sensor placement
* Any patients being monitored with motor evoked potential devices
* Any patients with a known hemoglobinopathy
* Any patients undergoing Cardio-Pulmonary Bypass (CPB)
* Any patients who cannot be transfused or has refused consent for a blood transfusion
* Patients who are moribund/salvage cases as determined by the participating anesthesiologist in charge of management of the patient in the operating room
* Patients being treated by any artificial oxygen carriers within 30 days of hospital stay
* Patients being managed outside of an operating room, or in operating room with conditions not conducive to perform and complete the study procedures (including use of the hemoglobin monitoring device)
* Patients younger than 18 years old
* Patients who are pregnant
* Any patients expected to receive transfusion preoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population in this study is defined at two levels: 1.Consenting eligible Anesthesiologists, and 2. Eligible patients under the case of the consenting eligible Anesthesiologist. Each level has its own eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-01 (Estimated); Study Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Number of allogeneic Red Blood Cells (RBC) units transfused intraoperatively | perioperative period untill the end of surgery

SECONDARY OUTCOMES:
Hospital stay treatment - Occurrence of any allogeneic RBC transfusions intraoperatively | From end of surgery until 30 days after surgery
Hospital stay treatment - Total number of allogeneic RBC units transfused perioperatively during hospital stay | From end of surgery until 30 days after surgery
Hospital stay treatment - Incidence of new (or worsening of pre-existing) ischemic events | From end of surgery until 30 days after surgery
Hospital stay treatment - 30-day mortality | From end of surgery until 30 days after surgery
Hospital stay treatment - Length of post-surgery hospital stay | From end of surgery until 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Idit Matot, professor, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel-Aviv Sourasky Medical Center, Tel Aviv, Israel